CLINICAL TRIAL: NCT02673944
Title: An Accuracy Study to Assess the Performance of the Peritron+ in Measuring Vesical Pressure in Patients in Comparison With Standard Urodynamic Measurements
Brief Title: Portable Pves Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PLUS-PVES-01
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peritron+ (Experimental): Patients will undergo a routine urodynamic evaluation, the Peritron+ will be used in conjunction with a water-based urodynamic catheter
  Interventions: Device: Peritron+

INTERVENTIONS:
Device: Peritron+ — Peritron+ will be connected to a standard urodynamic analyzer system to measure vesical pressure

SUMMARY:
A comparative study will be conducted and the patient will undergo a conventional urodynamic study. In order to successfully determine if the Peritron+ is capturing vesical pressure measurements consistent with conventional urodynamics the two sources of Pves will be collected concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Patients normally indicated for urodynamic evaluation

Exclusion Criteria:

* Patients who suffer from bladder infections
* Patients who suffer from strictures in the urethra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peritron+
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Peritron+
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Accurate Vesical PRessure
Description: To validate that the Peritron+ digital readings are identical to the urodynamic readings (+/- 3 cm H2O) in the sitting position.
Time Frame: During a routine urodynamic study (1 hr approx)
Measure: Mean (Standard Deviation); unit: cm H2O
Groups:
- Standard Urodynamic Analyzer: Patients will undergo a routine urodynamic evaluation, which will collect both Peritorn+ and UDS data.
Arm/Group | Peritron+ | Standard Urodynamic Analyzer
Number analyzed (Participants) | 10 | 10
cm H2O | 18.56 (8.29) | 17.45 (7.85)

ADVERSE EVENTS:
Arm/Group | Peritron+
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No